CLINICAL TRIAL: NCT00131131
Title: Epidemiology of Gallbladder Sludge & Stones in Pregnancy
Brief Title: Epidemiology of Gallbladder Sludge and Stones in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DK46890 (completed 2006); R01DK046890 (NIH)
Record Dates: First submitted 2005-08-16; First posted 2005-08-17 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Cholelithiasis
Keywords: physical activity; cholelithiasis; pregnancy complication
MeSH Terms: conditions — Cholelithiasis; Motor Activity; Pregnancy Complications | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): The intervention was an exercise program of moderate to vigorous intensity. The intervention started with 30-minute sessions three times per week, with the ultimate goal to have participants exercise four to five times per week for 45 to 60 minutes per session.
  Interventions: Behavioral: Exercise
- Control (No Intervention): Women in the control group did not attend instructional sessions with the exercise interventionist and did not receive the motivational mailings

INTERVENTIONS:
Behavioral: Exercise
  Arms: Exercise

SUMMARY:
The specific objective of this project is to study the impact exercise has on gallstone formation during pregnancy when women are at increased risk due to biochemical and physiological alterations.

DETAILED DESCRIPTION:
The female gender and multiparity are the two most important positive correlates of cholesterol gallstone disease. Pregnancy represents the period of time when the 'lithogenic' pressure on a woman is the highest. Biliary sludge is a precursor stage of gallstones. The investigators studied the etiological factors associated with the development of sludge and stones during pregnancy, and their early results suggest that it is inversely related to physical activity. They also found that being overweight, a known risk factor for gallstone disease, is associated with high blood leptin levels. In addition, the risk associated with high leptin levels is partially mitigated by physical activity.

In order to disentangle the effects of physical activity, leptin and gestational diabetes on gallbladder disease risk, and to understand the mechanisms behind the observed associations, the investigators propose to conduct a randomized controlled trial. This interventional study is a logical extension of their previous observational investigation. Their specific aims are:

* To evaluate whether an endurance exercise program is associated with lower risk of gallbladder disease in overweight pregnant women;
* To evaluate whether an endurance exercise intervention program changes leptin levels in pregnancy among overweight women;
* To examine the associations between gallbladder disease incidence and potential causal variables in this prospective trial. These variables include leptin levels, HDL, insulin levels, BMI (as it varies within women classified as overweight), as well as changes in these variables.

Gallstone disease affects 15-20% of adult Americans. Cholecystectomy is one of the most commonly performed operations. The morbidity, and the burden of cost, incurred by gallstones are staggering. Yet there is a dearth of understanding in the epidemiology and the cause of this disease. The results of this investigation should generate new, important and useful insights into the pathogenesis, and provide a rational strategy for the prevention, of this common and costly disease.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Over 18 years of age
* Eligible for care at Madigan Army Medical Center

Exclusion Criteria:

* Prior gallbladder surgery
* Non-English speaking
* Medical reason not to exercise during pregnancy
* Moving from area within 3 months

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1196 (Actual)
Dates: Start 2003-05; Primary Completion 2008-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Development of gall bladder sludge or gallstones | 18 and 36 weeks gestation
  Gallbladder sludge was defined as the presence of low amplitude echoes within the gallbladder without postacoustic shadowing, which could layer with positioning of the patient. Gallstones were defined as high amplitude echoes with postacoustic shadowing.

SECONDARY OUTCOMES:
Insulin | 18 and 36 weeks gestation
  Insulin, mU/mL
Leptin | 18 and 36 weeks gestation
  Leptin pg/L
Adiponectin | 18 and 36 weeks gestation
  Adiponectin pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Sum P Lee, MD, PhD, Principal Investigator — University of Washington; Shirley Beresford, PhD, Study Director — University of Washington School of Public Health and Community Medicine
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

REFERENCES:
- [Result] Ko CW, Napolitano PG, Lee SP, Schulte SD, Ciol MA, Beresford SA. Physical activity, maternal metabolic measures, and the incidence of gallbladder sludge or stones during pregnancy: a randomized trial. Am J Perinatol. 2014 Jan;31(1):39-48. doi: 10.1055/s-0033-1334455. Epub 2013 Mar 1. PMID 23456902